CLINICAL TRIAL: NCT02154126
Title: PRECISE: A Prospective, Multi-Center Evaluation of the Accuracy of a Novel Continuous Implanted Glucose Sensor
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0004
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accuracy assessment (Other)
  Interventions: Device: Continuous Glucose Monitoring Device (Senseonics)

INTERVENTIONS:
Device: Continuous Glucose Monitoring Device (Senseonics)

SUMMARY:
The purpose of this clinical investigation is to evaluate the accuracy of the Senseonics Continuous Glucose Monitoring System (Senseonics CGM System) measurements when compared with reference standard measurements (YSI glucose analyzer). The investigation will also evaluate safety of the Senseonics CGM System usage, while in the clinic and during home use.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following inclusion criteria will be included in this study:

1. Males and females ≥18 years of age
2. Clinically confirmed diagnosis of diabetes mellitus for a duration of 1 year and uses insulin therapy for their diabetes management (including subjects on insulin pump therapy)
3. Subject has signed an informed consent document and is willing to comply with protocol requirements

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be excluded from this study:

1. History of severe hypoglycemia in the last 6 months prior to study start, defined as hypoglycemia resulting in loss of consciousness or seizure
2. Diabetic ketoacidosis in the past 6 months
3. Any condition preventing or complicating the placement, operation or removal of the Sensor including upper extremity deformities or skin condition.
4. Any medical condition or illness that in the judgment of the investigator might interfere with the procedures, results or compliance during the course of this investigation, or increase the risk of induced hypoglycemia or repeated blood testing including significantly impaired hepatic function and renal failure
5. Known microvascular (diabetic) complications, including active proliferative diabetic retinopathy or macular edema, active non-proliferative retinopathy, diabetic nephropathy including active retinopathy
6. Hematocrit >50% or <30%
7. Females lactating or pregnant or intending to become pregnant during the course of the investigation
8. A condition requiring or likely to require magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Accuracy (mean absolute relative difference) compared to be reference device should be less than 20% | 90 days
  To determine accuracy of the Senseonics CGM System measurements over successive periods of 30 days of Sensor use through 180 days post-insertion.

CONTACTS AND LOCATIONS:
Overall Officials: J.Hans de Vries, MD, Principal Investigator — Academic Medical Centre
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands

REFERENCES:
- [Derived] Kropff J, Choudhary P, Neupane S, Barnard K, Bain SC, Kapitza C, Forst T, Link M, Dehennis A, DeVries JH. Accuracy and Longevity of an Implantable Continuous Glucose Sensor in the PRECISE Study: A 180-Day, Prospective, Multicenter, Pivotal Trial. Diabetes Care. 2017 Jan;40(1):63-68. doi: 10.2337/dc16-1525. Epub 2016 Nov 4. PMID 27815290